CLINICAL TRIAL: NCT03625037
Title: A Phase 1/2, Open-label Safety Trial of GEN3013 in Patients With Relapsed, Progressive or Refractory B-Cell Lymphoma
Brief Title: First-in-Human (FIH) Trial in Patients With Relapsed, Progressive or Refractory B-Cell Lymphoma
Acronym: EPCORE™ NHL-1
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Genmab (Industry)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GCT3013-01; 2017-001748-36 (EudraCT Number); NL64317.078.17 (Registry Identifier: CCMO); 241053 (Other: IRAS ID; UK Research Summaries Database); 2023-504802-12-00 (EU CTIS Number)
Expanded Access: NCT05733650 (Approved for marketing)
Record Dates: First submitted 2018-06-07; First posted 2018-08-10 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: DLBCL; High-grade B-cell Lymphoma (HGBCL); Primary Mediastinal Large B-cell Lymphoma (PMBCL); FL; MCL; Small Lymphocytic Lymphoma (SLL); Marginal Zone Lymphoma (MZL); Indolent B-cell Non-Hodgkin Lymphoma (iNHL); Aggressive B-cell Non-Hodgkin Lymphoma (aNHL)
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, B-Cell, Marginal Zone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Epcoritamab (Experimental): Epcoritamab will be administered by subcutaneous injections in cycles of 28 days.
  Interventions: Biological: Epcoritamab

INTERVENTIONS:
Biological: Epcoritamab — Administered as specified in the treatment arm.
  Other Names: GEN3013; DuoBody®-CD3xCD20; EPKINLY™

SUMMARY:
The purpose of this trial is to measure the following in participants with relapsed and/or refractory B-cell lymphoma who receive epcoritamab, an antibody also known as EPKINLY™ and GEN3013 (DuoBody®-CD3xCD20):

* The dose schedule for epcoritamab
* The side effects seen with epcoritamab
* What the body does with epcoritamab once it is administered
* What epcoritamab does to the body once it is administered
* How well epcoritamab works against relapsed and/or refractory B-cell lymphoma

The trial consists of 3 parts:

* a dose-escalation part (Phase 1, first-in-human [FIH])
* an expansion part (Phase 2a)
* a dose-optimization part (OPT) (Phase 2a)

The trial time for each participant depends on which trial part the participant enters:

* For the dose-escalation part, each participant will be in the trial for approximately 1 year, which is made up of 21 days of screening, 6 months of treatment (the total time of treatment may be different for each participant), and 6 months of follow-up (the total time of follow-up may be different for each participant).
* For the expansion and dose-OPT parts, each participant will be in the trial for approximately 1.5 years, which is made up of 21 days of screening, 1 year of treatment (the total time of treatment may be different for each participant), and 6 months of follow-up (the total time of follow-up may be different for each participant).

Participation in the study will require visits to the sites. During the first month, participants must visit every day or every few days, depending on which trial part the participant enters. After that, participants must visit weekly, every other week, once a month, and once every 2 months, as trial participation ends.

All participants will receive active drug, and no participants will be given placebo.

DETAILED DESCRIPTION:
The purpose of the dose-escalation part of the trial is to determine the maximum tolerated dose (MTD) and the recommended Phase 2 dose (RP2D), as well as to establish the safety profile of epcoritamab in participants with relapsed or refractory B-cell lymphoma.

In the expansion part, additional participants will be treated with epcoritamab, at the RP2D and the purpose is to further explore and determine the safety and efficacy of epcoritamab.

The dose-OPT part will evaluate alternative priming and intermediate dose regimens of epcoritamab in participants with:

* Diffuse large B-cell lymphoma (DLBCL)
* Follicular lymphoma (FL)
* Mantle cell lymphoma (MCL)

All participants will receive epcoritamab at the RP2D.

ELIGIBILITY:
Main Inclusion Criteria - Escalation Part (recruitment completed)

* Documented CD20+ mature B-cell neoplasm

  1. DLBCL - de novo or transformed
  2. HGBCL
  3. PMBCL
  4. FL
  5. MCL
  6. SLL
  7. MZL (nodal, extranodal or mucosa associated)
* Relapsed and/or refractory disease following treatment with an anti-CD20 monoclonal antibody (e.g. rituximab) potentially in combination with chemotherapy and/or relapsed after autologous stem cell rescue.
* Eastern Cooperative Oncology Group (ECOG) performance status 0,1 or 2.
* Participants must have measurable disease by computed tomography (CT), magnetic resonance imaging (MRI) or Positron emission tomography-Computed tomography (PET-CT) scan
* Acceptable renal function.
* Acceptable liver function.

Main Inclusion Criteria - Expansion & Dose-OPT Parts

* Documented CD20 positive mature B cell neoplasm or CD20+ MCL.
* DLBCL, de novo or transformed (including double hit or triple hit).
* PMBCL
* FL grade 3B
* Histologic confirmed FL
* MZL
* SLL
* MCL (prior Bruton's tyrosine kinase inhibitor [BTKi] or intolerant to BTKi)
* At least 2 therapies including an anti-CD20 monoclonal antibody containing chemotherapy combination regimen.
* Either failed prior autologous hematopoietic stem cell transplantation (HSCT) or ineligible for autologous stem cell transplantation due to age or comorbidities.
* At least 1 measurable site of disease based on CT, MRI or PET-CT scan with involvement of 2 or more clearly demarcated lesions and or nodes.

Main Exclusion Criteria - All Parts

* Primary central nervous system (CNS) lymphoma or CNS involvement by lymphoma at screening.
* Known past or current malignancy other than inclusion diagnosis.
* Aspartate aminotransferase (AST), and/or alanine transaminase (ALT) >3 × upper limit of normal.
* Total bilirubin >1.5 × upper limit of normal, unless bilirubin rise is due to Gilbert's syndrome or of non-hepatic origin.
* Estimated Creatinine clearance (CrCl) <45 milliliters (mL)/min.
* Known clinically significant cardiovascular disease.
* Ongoing active bacterial, viral, fungal, mycobacterial, parasitic, or other infection requiring systemic treatment (excluding prophylactic treatment). Past coronavirus disease 2019 (COVID-19) infection may be a risk factor.
* Confirmed history or current autoimmune disease or other diseases resulting in permanent immunosuppression or requiring permanent immunosuppressive therapy.
* Seizure disorder requiring therapy (such as steroids or anti-epileptics).
* Any prior therapy with an investigational bispecific antibody targeting CD3 and CD20.
* Prior treatment with chimeric antigen receptor T-cell (CAR-T) therapy within 30 days prior to first epcoritamab administration.
* Eligible for curative intensive salvage therapy followed by high dose chemotherapy with HSCT rescue.
* Autologous HSCT within 100 days prior to first epcoritamab administration, or any prior allogeneic HSCT or solid organ transplantation.
* Active hepatitis B (deoxyribonucleic acid [DNA] polymerase chain reaction [PCR]-positive) or hepatitis C (ribonucleic acid [RNA] PCR-positive infection). Participants with evidence of prior hepatitis B (HBV) but who are PCR-negative are permitted in
* Known human immunodeficiency virus (HIV) infection.
* Exposed to live or live attenuated vaccine within 4 weeks prior to signing Informed consent form (ICF).
* Pregnancy or breast feeding.
* Participant is known or suspected of not being able to comply with the study protocol or has any condition for which, participation would not be in the best interest of the participant.
* Contraindication to all uric acid lowering agents.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 666 (Actual)
Dates: Start 2018-06-26 (Actual); Primary Completion 2029-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Dose-Escalation: Dose Limiting Toxicity (DLT) | During the first cycle (28 days)
  To determine the MTD and/or RP2D to be studied in the Expansion part. DLT will be graded according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0.
Dose-Escalation: Number of Participants with Adverse Events (AEs) | From first dose until the end of the safety follow-up period (Up to 1 year)
  An AE is any untoward medical occurrence in a clinical trial participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product.
Expansion: Overall Response Rate (ORR) | Up to 1.5 years
  ORR is defined as the percentage of participants achieving complete response (CR) or partial response (PR) based on Lugano criteria.
Dose-OPT DLBCL, FL and MCL: Percentage of Participants with =>Grade 2 Cytokine Release Syndrome (CRS) Events and All Grade CRS Events | From first dose until 7 days after second full dose (Day 28 for DLBCL; Day 35 for FL; Day 28-35 for MCL)
  CRS will be graded based on American Society for Transplantation and Cellular Therapy (ASTCT) criteria.

SECONDARY OUTCOMES:
Dose-Escalation: Number of Participants with Anti-lymphoma Activity of Epcoritamab | Up to 1 year
  Anti-lymphoma activity will be evaluated as number of participants with resolution of constitutional symptoms, reduction in tumor size, objective, and best response (ORR, CR and PR).
Dose-Escalation: Duration of Response (DOR) | Up to 1 year
  DOR is defined as the time from the first documentation of response (CR or PR) to the date of progressive disease (PD) or death, whichever occurs earlier as assessed by the investigator.
Expansion: DOR | Up to 1.5 years
  DOR is defined as the time from the first documentation of response (CR or PR) to the date of PD or death, whichever occurs earlier based on Lugano criteria.
Expansion Part: Changes in Lymphoma Symptoms as Measured by the Functional Assessment of Cancer Therapy - Lymphoma (FACT-Lym) | Up to 1.5 year
  Change from baseline in health-related quality of life over time and in relation to treatment will be evaluated using FACT-Lym scale.
Dose-OPT DLBCL and FL: Percentage of Participants with >=Grade 2 CRS Events and All Grade CRS Events Following First Full Dose | Up to 1.5 years
  CRS will be graded based on ASTCT criteria.
Dose-OPT DLBCL and FL: Percentage of Participants with >=Grade 2 CRS Events and All Grade CRS Events Overall | Up to 1.5 years
  CRS will be graded based on ASTCT criteria.
Dose-OPT DLBCL and FL: ORR | Up to 1.5 years
  ORR is defined as the percentage of participants achieving CR or PR assessed by investigator.
Dose-OPT DLBCL and FL: CR Rate | Up to 1.5 years
  CR rate is defined as the percentage of participants with CR assessed by investigator.
Dose-OPT DLBCL and FL: Duration of CR (DoCR) | Up to 1.5 years
  DoCR is defined as the time from the first documentation of CR to the date of PD or death, whichever occurs earlier assessed by investigator.
Dose-OPT DLBCL and FL: Progression-Free Survival (PFS) | Up to 1.5 years
  PFS is defined as the time from Day 1 of Cycle 1 to first documented PD or death due to any cause, whichever occurs earlier assessed by investigator.
Dose-OPT DLBCL and FL: DLT | During the first cycle (28 days) in each Dose-OPT Part (DLBCL, FL and MCL)
  To determine the MTD and/or RP2D to be studied in the expansion part. DLT will be graded according to NCI-CTCAE version 5.0.
Dose-OPT DLBCL, FL and MCL: DOR | Up to 1.5 years
  DOR is defined as the time from the first documentation of response (CR or PR) to the date of PD or death, whichever occurs earlier based on Lugano criteria assessed by investigator.
Dose-Escalation and Dose-OPT DLBCL, FL and MCL: Pre-dose Values of Epcoritamab | Predose and postdose at multiple timepoints of each Cycle (Cycle length=28 days), up to approximately 1.5 years
Dose-Escalation, Expansion Part and Dose-OPT MCL: PFS | Dose-Escalation: Up to 1 year; Expansion and Dose-OPT Part (MCL): 1.5 years
  PFS is defined as the time from Day 1 of Cycle 1 to first documented PD or death due to any cause, whichever occurs earlier based on Lugano criteria.
Expansion and Dose-OPT MCL: CR Rate | Up to 1.5 years
  CR rate is defined as the percentage of participants with CR based on Lugano criteria.
Expansion and Dose-OPT MCL: DoCR | Up to 1.5 years
  DoCR is defined as the time from the first documentation of CR to the date of PD or death, whichever occurs earlier based on Lugano criteria.
Expansion and Dose-OPT MCL: ORR | Up to 1.5 years
  ORR is defined as the percentage of participants achieving CR or PR based on LYRIC.
Expansion: Time to Response (TTR) | Up to 1.5 years
  TTR is defined as the time from Day 1 of Cycle 1 to first documentation of objective tumor response (PR or better) earlier based on Lugano criteria.
Expansion and Dose-OPT MCL: CR Rate | Up to 1.5 years
  CR rate is defined as the percentage of participants with CR based on LYRIC.
Expansion and Dose-OPT MCL: PFS | Up to 1.5 years
  PFS is defined as the time from Day 1 of Cycle 1 to first documented PD or death due to any cause, whichever occurs earlier based on LYRIC.
Expansion and Dose-OPT MCL: DOR | Up to 1.5 years
  DOR is defined as the time from the first documentation of response (CR or PR) to the date of PD or death, whichever occurs earlier based on LYRIC.
Expansion and Dose-OPT MCL: DoCR | Up to 1.5 years
  DoCR is defined as the time from the first documentation of CR to the date of PD or death, whichever occurs earlier based on LYRIC.
Expansion and Dose-OPT: TTR | Up to 1.5 years
  TTR is defined as the time from Day 1 of Cycle 1 to first documentation of objective tumor response (PR or better) earlier based on LYRIC.
Expansion and Dose-OPT DLBCL, FL and MCL: Number of Participants with AEs | Up to 7 years and 6 months
  An AE is any untoward medical occurrence in a clinical trial participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product.
Expansion and Dose-OPT DLBCL, FL and MCL: Rate of Minimal Residual Disease (MRD) Negativity | Up to 1.5 years
  MRD is defined as percentage of participants with at least 1 MRD negative result.
All Parts: Number of Participants with CRS Events | Up to Day 1 of Cycle 12 (Cycle length=28 days)
  CRS will be graded based on ASTCT criteria.
All Parts: Total Body Clearance of Epcoritamab from the Plasma (CL) | Predose and postdose at multiple timepoints of each cycle (Cycle length=28 days), Dose-Escalation: Up to 1 year; Expansion and Dose-OPT Part: Up to 1.5 years
All Parts: Area under Curve (AUC) of Epcoritamab | Predose and postdose at multiple timepoints of each cycle (Cycle length=28 days), Dose-Escalation: Up to 1 year; Expansion and Dose-OPT Part: Up to 1.5 years
All Parts: Maximum (peak) Plasma Concentration (Cmax) of Epcoritamab | Predose and postdose at multiple timepoints of each cycle (Cycle length=28 days), Dose-Escalation: Up to 1 year; Expansion and Dose-OPT Part: Up to 1.5 years
All Parts: Time to Reach Cmax of Epcoritamab | Predose and postdose at multiple timepoints of each cycle (Cycle length=28 days), Dose-Escalation: Up to 1 year; Expansion and Dose-OPT Part: Up to 1.5 years
All Parts: Half Life of Epcoritamab (t1/2) | Predose and postdose at multiple timepoints of each cycle (Cycle length=28 days), Dose-Escalation: Up to 1 year; Expansion and Dose-OPT Part: Up to 1.5 years
All Parts: Number of Participants with Anti-drug Antibody (ADA) | Up to 7 years and 6 months
  Plasma samples will be screened for antibodies binding to epcoritamab, and for confirmed positive samples, the titer against the two specific arms of epcoritamab will be reported.
All Parts: Time to Next Anti-lymphoma Therapy (TTNT) | Dose-Escalation: Up to 1 year; Expansion and Dose-OPT Part (DLBCL, FL and MCL): Up to 1.5 years
  TTNT is defined as the time from Day 1 of Cycle 1 to first recorded administration of subsequent anti-lymphoma therapy or death due to any cause, whichever occurs earlier.
All Parts: Overall survival (OS) | Dose-Escalation: Up to 1 year; Expansion and Dose-OPT Part DLBCL, FL and MCL: Up to 1.5 years
  OS is defined as the time from Day 1 of Cycle 1 to death.
Expansion: Trough Concentration of Epcoritamab | Up to 1.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Study Official, Study Director — Genmab
Locations (85):
- United States (17):
  - Arizona Mayo Clinic, Phoenix, Arizona
  - University of California at San Francisco, San Francisco, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - University of Iowa Hospital and Clinics, Iowa City, Iowa
  - Ochsner Medical Center, New Orleans, Louisiana
  - University of Michigan, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Hackensack Meridian Health, Hackensack, New Jersey
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - OHSU Knight Cancer Institute, Portland, Oregon
  - Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - UT Southwestern, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
- Australia (10):
  - Monash Health, Clayton
  - Concord Hospital, Concord
  - St. Vincent Hospital, Fitzroy
  - Royal Brisbane and Women's Hospital, Herston
  - Royal Hobart Hospital RHH, Hobart
  - St. George Hospital, Kogarah
  - Cabrini Hospital, Malvern
  - Sir Charles Gairdner Hospital, Nedlands
  - Gold Coast Hospital, Southport
  - Westmead Hospital, Sydney
- Canada (2):
  - Tom Baker Cancer Care, Calgary
  - Toronto-Sunnybrook Regional Cancer Ctr, Toronto
- Denmark (3):
  - Rigshospitalet, Copenhagen
  - Odense University Hospital, Odense
  - Vejle Hospital, Vejle
- Finland (3):
  - Helsinki University Hospital, Helsinki
  - Kuopio University Hospital, Kuopio
  - Tampere University Hospital, Tampere
- France (6):
  - Hopital Henri Mondor, Créteil
  - CHU Montpellier, Montpellier
  - Hospital Saint-Louis, Paris
  - Hospices Civils de Lyon Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Centre Henri Becquerel, Rouen
  - CHU de Tours-Hopital Bretonneau, Tours
- Germany (6):
  - Charite - Universitaetsmedizin Berlin, Berlin
  - Klinik fur Innere Medizin Hamatologie and Onkologie, Berlin
  - Universitaetsklinikum Koeln, Cologne
  - Universitaetsklinikum Essen, Essen
  - Johannes Gutenberg University, Mainz
  - Der Universität Munchen Medizinische Klinik III LMU, München
- Italy (5):
  - Ao Ss Antonio E Biagio Alessandria, Alessandria
  - Policlinico S. Orsola-Ematologia LA Seragnoli, Bologna
  - Istituto di Candiolo- Fondazione del Piemonte per l'Oncologia, Candiolo
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori, Meldola
  - IRCCS Ospedale San Raffaele, Milan
- Netherlands (4):
  - VU University Medical Center, Amsterdam
  - Maastricht University Medical Center, Maastricht
  - Erasmus MC Cancer Institute, Rotterdam
  - Universitair Medisch Centrum Utrecht, Utrecht
- Poland (6):
  - Szpital Uniwersytecki nr 2 im dr. Jana Biziela, Bydgoszcz
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Pratia-McM, Krakow
  - Wojewodzki Szpital Specjalistyczny im. Janusza Korczaka, Słupsk
  - Maria Sklodowska-Curie Memorial Cancer Center and Institute, Warsaw
  - Uniwersytecki Szpital Kliniczny im. Jana Mikulicza-Radeckiego, Wroclaw
- Singapore (2):
  - National University Hospital, Singapore
  - Singapore General Hospital, Singapore
- South Korea (9):
  - Dong-A University Hospital, Busan
  - Keimyung University Dongsan Medical Center, Daegu
  - National Cancer Center, Goyang-si
  - Chonbuk National University Hospital, Jeonju
  - Seoul National University Bundang Hospital, Seongnam-si
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University, Seoul
- Spain (5):
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - Hospital Germans Trias i Pujol, Badalona
  - Hospital Universitario Vall dHebron, Barcelona
  - Institut Catala de Oncologia, Barcelona
  - Hospital Universitario Fundacin Jimnez Daz, Madrid
- Sweden (3):
  - Skåne University Hospital, Lund
  - Karolinska University Hospital Huddinge, Stockholm
  - Akademiska sjukhuset Uppsala University Hospital, Uppsala
- United Kingdom (4):
  - The Christie NHS Foundation Trust, Manchester
  - Plymouth University School of Medicine- Derriford Hospital, Plymouth
  - University Hospital Southampton NHS Foundation Trust, Southampton
  - Royal Marsden NHS Foundation Trust, Sutton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Thieblemont C, Phillips T, Ghesquieres H, Cheah CY, Clausen MR, Cunningham D, Do YR, Feldman T, Gasiorowski R, Jurczak W, Kim TM, Lewis DJ, van der Poel M, Poon ML, Cota Stirner M, Kilavuz N, Chiu C, Chen M, Sacchi M, Elliott B, Ahmadi T, Hutchings M, Lugtenburg PJ. Epcoritamab, a Novel, Subcutaneous CD3xCD20 Bispecific T-Cell-Engaging Antibody, in Relapsed or Refractory Large B-Cell Lymphoma: Dose Expansion in a Phase I/II Trial. J Clin Oncol. 2023 Apr 20;41(12):2238-2247. doi: 10.1200/JCO.22.01725. Epub 2022 Dec 22. PMID 36548927
- [Result] Linton KM, Vitolo U, Jurczak W, Lugtenburg PJ, Gyan E, Sureda A, Christensen JH, Hess B, Tilly H, Cordoba R, Lewis DJ, Okada C, Hutchings M, Clausen MR, Sancho JM, Cochrane T, Leppa S, Chamuleau MED, Gernhardt D, Altintas I, Liu Y, Ahmadi T, Dinh MH, Hoehn D, Favaro E, Elliott B, Thieblemont C, Vose JM. Epcoritamab monotherapy in patients with relapsed or refractory follicular lymphoma (EPCORE NHL-1): a phase 2 cohort of a single-arm, multicentre study. Lancet Haematol. 2024 Aug;11(8):e593-e605. doi: 10.1016/S2352-3026(24)00166-2. Epub 2024 Jun 15. PMID 38889737
- [Derived] Danilov AV, Kambhampati Thiruvengadam S, Linton K, Cumings K, Chirikov V, Mutebi A, Bains Chawla S, Chhibber A, Rivas Navarro F, Marques Goncalves F, Wang A, Ding Z, Alshreef A, Favaro E, Hoehn D, Sureda A. Indirect comparison of epcoritamab vs chemoimmunotherapy, mosunetuzumab, or odronextamab in follicular lymphoma. Blood Adv. 2025 Aug 12;9(15):3754-3765. doi: 10.1182/bloodadvances.2024015274. PMID 40472301
- [Derived] Thieblemont C, Karimi YH, Ghesquieres H, Cheah CY, Clausen MR, Cunningham D, Jurczak W, Do YR, Gasiorowski R, Lewis DJ, Kim TM, van der Poel M, Poon ML, Feldman T, Linton KM, Sureda A, Hutchings M, Dinh MH, Kilavuz N, Soong D, Mark T, Sacchi M, Phillips T, Lugtenburg PJ. Epcoritamab in relapsed/refractory large B-cell lymphoma: 2-year follow-up from the pivotal EPCORE NHL-1 trial. Leukemia. 2024 Dec;38(12):2653-2662. doi: 10.1038/s41375-024-02410-8. Epub 2024 Sep 25. PMID 39322711
- [Derived] Phillips T, Lugtenburg P, Kalsekar A, Mutebi A, Wang A, Blaedel J, Kosa K, Martin S, Sacchi M, Kilavuz N, Thieblemont C. Improvements in Patient-Reported Outcomes in Relapsed or Refractory Large B-Cell Lymphoma Patients Treated With Epcoritamab. Clin Lymphoma Myeloma Leuk. 2024 Mar;24(3):e78-e87.e2. doi: 10.1016/j.clml.2023.11.005. Epub 2023 Nov 27. PMID 38151388
- [Derived] Hutchings M, Mous R, Clausen MR, Johnson P, Linton KM, Chamuleau MED, Lewis DJ, Sureda Balari A, Cunningham D, Oliveri RS, Elliott B, DeMarco D, Azaryan A, Chiu C, Li T, Chen KM, Ahmadi T, Lugtenburg PJ. Dose escalation of subcutaneous epcoritamab in patients with relapsed or refractory B-cell non-Hodgkin lymphoma: an open-label, phase 1/2 study. Lancet. 2021 Sep 25;398(10306):1157-1169. doi: 10.1016/S0140-6736(21)00889-8. Epub 2021 Sep 8. PMID 34508654